CLINICAL TRIAL: NCT01506219
Title: Geriatrician-performed Comprehensive Geriatric Care in Older Adults Referred to an Outpatient Community Rehabilitation Unit
Brief Title: Geriatrician-performed Comprehensive Geriatric Care in an Outpatient Community Rehabilitation Unit
Acronym: GCGCCRU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NZ-151111-VHDZ
Record Dates: First submitted 2011-12-28; First posted 2012-01-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-10

CONDITIONS: Fragility
Keywords: Randomized controlled trial; Comprehensive geriatric care; Activity of daily living; Quality of life; Healthcare utilization; Community rehabilitation unit; Medication adjustment

STUDY DESIGN:
Intervention Model Description: A pragmatic open assessor-blinded clinical randomized controlled trial with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: The geriatrician was blinded to the primary endpoint data that were drawn from the National Patient Registry via Researcher Service. The dataset was generated by the Registry's staff blinded to the patient allocation.
  It was impossible to blind the participants and their relatives or the geriatrician and the rehabilitation units' staff to the allocation group.
  The research nurse was not blinded to patient allocation for practical reasons. The research occupational therapist was blinded to treatment allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Geriatrician-performed CGC (Experimental): Geriatrician-performed CGC in addition to the usual care at Community Rehabilitation Unit.
  Interventions: Procedure: Geriatrician-performed CGC
- Usual care (No Intervention): Usual services at Community Rehabilitation Unit.

INTERVENTIONS:
Procedure: Geriatrician-performed CGC — Individual disease management and coping was provided using the holistic approach during the face-to-face counselling, where the actual problems, expectations and aims were defined in dialogue with the patient and/or relatives. Afterwards, targeted problem solving with focus on the potentially reversible causes of functional deterioration was established. Finally, medication adjustment was carried out with particular attention to drugs which may lead to iatrogenic functional deterioration, delirium, falls, and malnutrition. Furthermore, the intervention included intravenous antibiotics or blood transfusions (if indicated) conducted by the geriatrician at the rehabilitation units.
  Arms: Geriatrician-performed CGC

SUMMARY:
Introduction:

Older adults with multiple illnesses represent the fastest growing sector of society and make increasing demands on all sectors of the health care system, particularly in outpatient community rehabilitation units due to shorter time of stay in acute care units and hospitals. The aim of this study is to investigate the effect of geriatrician-performed comprehensive geriatric care (CGC) in older people referred to an outpatient community rehabilitation unit.

Methods:

The study is a prospective randomized controlled trial. Settings: two community care rehabilitation units in Aarhus Municipality, Denmark. Inclusion: persons aged 65 and older from home or hospital. Exclusion: persons who received palliative care or had been assessed by a geriatrician during the past month. Intervention: medical history, physical examination, blood tests, medication adjustment and related treatments performed by a geriatrician. Control: usual care in a community rehabilitation unit. Number of hospital admissions and emergency department (ED) visits (primary outcome), number of GP contacts, activities of daily living, physical and cognitive functioning, quality of life, data on institutionalization, medication status, and mortality are assessed at day 30 and 90 after arrival at the rehabilitation unit.

Project status:

The outpatient CGC model is developed, implemented and compared with usual care in a pragmatic RCT.

DETAILED DESCRIPTION:
Procedure Participants were recruited consecutively from the rehabilitation unit Vikaergaarden in the period from January 17, 2012 to May 29, 2015, and from the rehabilitation unit Thorsgaarden from October 20, 2014 to May 29, 2015. The random allocation of the participants to an intervention group (IG) or a control group (CG) was done by an independent external organization ("TrialPartner", Public Health and Quality Improvement, Central Denmark Region). The permuted block sizes stratified the randomization according to sex, age, and place of referral. The randomization took place within three days after the participants' arrival to the rehabilitation unit. Owing to the nature of this study, it was impossible to blind participants and their relatives to the allocation group. The project manager was blinded to the study outcomes, which were collected from the registers or by the blinded research occupational therapist. Rehabilitation units' staff, particularly physiotherapists, were not blinded.

Care in the CG The patients were referred for rehabilitation either from hospital or home by the hospital personnel or by the home care staff.The typical standard rehabilitation and care program lasts five weeks. The interdisciplinary approach is based on the patient's whole situation, capability and wishes/needs. On the first day of rehabilitation, the patient's functional status is observed by the rehabilitation unit's physiotherapists and occupational therapists, and a nutritional screening is performed by the rehabilitation unit's nutritionist.The team members discuss the patient's discharge destination and necessary arrangements with the patient and his/her relatives at the mid-term meeting and before discharge from the rehabilitation unit. Municipality nurse participates in these meeting personally or by telephone. Destination after discharge is based upon the patient's motivation, functional and medical status.

The patient's GPs visit the patients during the stay if required or occasionally by own initiative depending on practice routine and geographical distance. GPs mostly visit frail and high-risk elderly patients especially if recently hospitalized. Acute medical aid is called for in case of illness after 4.p.m. and on weekends and public holidays.

Care in the IG Participants in the IG had the same access to usual care and additionally underwent a CGC performed by a physician specialized in geriatric medicine. The intervention included medical history, physical examination, blood tests, medication adjustment and treatments, including intravenous antibiotics or blood transfusions conducted by the geriatrician at the rehabilitation units. The geriatrician was employed 18.5 hours per week and was present at the rehabilitation units for four days a week, and could be contacted on telephone for any reason by participants, their relatives, or the units' staff on weekdays from 8 a.m. to 3 p.m.

BaselineAssessments Before randomization baseline characteristics were registered from medical records by the project manager, comprising age, gender, place of referral, marital status, residence, previous diagnoses, list of medications and comorbidity burden by Charlson Comorbidity Index (CCI). Baseline functional status and quality of life measures were assessed on day 3 from admission to the rehabilitation units by a research occupational therapist.

Statistics The numbers of hospital admissions, ED visits, ambulatory contacts, and GP contacts will be compared by Incidence Rate Ratios (IRR) with 95% confidence intervals (CI). IRR will be calculated using negative binominal regression with adjustment for mortality by including the risk time as an exposure variable.

Mortality rates after 30 and 90 days will be calculated as percentages of deaths in total population per group. In non-survivors and in case of missing baseline observations, the missing measures will be set to the worst possible values. The worst value imputation method will be used in all other cases of missing values.

The mean group values will be analyzed using repeated measurements mixed model. Dichotomous variables will be created to investigate distribution between participants who worsened/did not change versus participants who improved their functional status or quality of life, and analyzed using logistic regression. Results will be expressed as odds ratios (ORs) with 95% CIs.

Subgroup analyses will be conducted to explore if effects of intervention when compared to usual care depended on the baseline comorbidity burden low/moderate (CCI 0-2) versus high (CCI ≥3 points). The subgroup analyses will be carried out for the functional status and quality of life.

There were no drop-outs during the study and data on healthcare utilization are complete. Intention-to-treat analyses will be performed in the all 368 participants. The two-sided significance level of 5% will be used for evaluation of statistical significance in the primary and secondary endpoints.

(The materials and methods are described in detail elsewhere: Zintchouk D, Lauritzen T, Damsgaard EM. "Comprehensive Geriatric Care Versus Standard Care For Elderly Referred To A Rehabilitation Unit - A Randomized Controlled Trial". J Aging Res Clin Practice 2017;inpress. Published online December 15, 2016, http://dx.doi.org/10.14283/jarcp.2016.126).

ELIGIBILITY:
Inclusion Criteria:

1. Age 65+ years old in Aarhus Municipality, Denmark
2. Referral to a community rehabilitation unit by general practitioner, home care services or a hospital department staff
3. Written informed consent

Exclusion Criteria:

1. Persons, who received Comprehensive Geriatric Assessment within last 1 month
2. Persons in the palliative care at the time of referral

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 368 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Number of hospital admissions and ED visits (the secondary healthcare utilization) | At 90 days after admission to the rehabilitation units
  Numbers of all hospital admissions and ED visits

SECONDARY OUTCOMES:
Number of ambulatory contacts (the secondary healthcare utilization) | At 90 days after admission to the rehabilitation unit (during + after the rehabilitation stay)
  All ambulatory contacts, except to the Department of Radiology
Number of days in hospital (the secondary healthcare utilization) | At 90 days after admission to the rehabilitation unit
  All days spent in hospital
Number of GP contacts (the primary healthcare utilization) | At 90 days after admission to the rehabilitation unit (during + after the rehabilitation stay)
  Numbers of all out of hour GP visits or phone calls, daytime GP consultations and visits, phone and email consultations, and other GP services
Mortality | At 30 and 90 days after admission to the rehabilitation unit.
  Mortality rates calculated as the percentage of deaths in the total population per Group (Cox regression analysis used to calculate hazard ratios)
Changes in ADL measured by the Modified Barthel-100 Index (MBI) | From the baseline assessment at day 3 to 10, 30 and 90 days after admission to the rehabilitation unit
  MBI is a 10-item instrument that provides a score of basic daily activities. The scores range from 0-100, with a higher score indicating greater independence. The MBI changes calculated as the mean differences in the MBI sum-scores, and as percentage of participants who worsened/did not change vs who improved their MBI from day 3 to day 90
Changes in Overall Quality of Life (OQoL) measured by the Depression List (DL). | From the baseline assessment at dag 3 to 10, 30 and 90 days after admission to the rehabilitation unit
  DL is an interview-based questionnaire validated among nursing home residents and can be completed by persons themselves with a MMSE score ≥ 5. DL consists of 15 questions covering emotional well-being, social relationships, life-satisfaction, comfort, functional competence, and autonomy. The scale ranges from 0 (best quality of life) to score 30 (poorest quality of life). DL changes calculated as the mean differences in the DL sum-scores, and as percentage of participants who worsened/did not change vs who improved their DL from day 3 to day 90
Changes in cognitive functioning measured by the Mini-mental state examenation (MMSE) | From the baseline assessment at dag 3 to 10, 30 and 90 days after admission to the rehabilitation unit
  MMSE is a 10-minute bedside measure of impaired thinking. The items of the MMSE include tests of orientation, registration, recall, calculation and attention, naming, repetition, comprehension, reading, writing and drawing.The MMSE changes calculated as the mean differences in the MMSE sum-scores, and as percentage of participants who worsened/did not change vs who improved their MMSE from day 3 to day 90
Changes in physical functioning measured by the 30-second Chair Stand Test (30s-CST) | From the baseline assessment at dag 3 to 10, 30 and 90 days after admission to the rehabilitation unit
  The 30-second chair stand test measures body strength, by determining the number of times the participant can stand up fully and sit down in 30 seconds, with the arms crossed over the chest. We have used the modified version of this test, where use of armrest is allowed. The 30-second Chair Stand Test changes calculated as the mean differences in the 30s-CST sum-scores, and as percentage of participants who worsened/did not change vs who improved their 30s-CST from day 3 to day 90
Residential status | Between baseline and 90 after admission to the rehabilitation unit
  Calculated in survivors as percentages of persons living in their own home, sheltered housing or nursing home
Walking aids use | Between baseline and 90 days after admission to the rehabilitation unit
  Percentages of participants using stick, walker or wheelchair
Personal social services extent | Between baseline and 90 days after admission to the rehabilitation unit
  Percentages of participants with the personal social services (included practical help and shopping, transport, and emergency call)
Home care | Between baseline and 90 days after admission to the rehabilitation unit
  Data on homecare in own home/sheltered housing obtained in survivors living in own home/sheltered housing, and calculated as percentages of persons with homecare (weekly or one or more times daily)
District nurses availability | Between baseline and 90 days after admission to the rehabilitation unit
  Data on district nurse availability in own home/sheltered housing obtained in survivors living in own home/sheltered housing, and calculated as percentages of persons with district nurses availability
Medication status and medication burden | Between baseline and 90 days after admission to the rehabilitation unit
  Calculated as percentages of the persons using regularly drugs according to their ATC codes. Polypharmacy was categorized into 3 groups based on the number of regular drugs prescribed. Hyper-polypharmacy was defined as concurrent prescription of 10 or more drugs per day; polypharmacy was defined as prescription of 5 to 9 drugs, and non-polypharmacy represented patients prescribed 4 or fewer drugs concomitantly. Medication burden were assessed in a pragmatic way by selection of specific medications with anticholinergic effects and sedative effects. The chose of the selected drugs matched the drugs where the indication should reassess in the older adults according to the National Board of Health.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Zintchouk, MD, Principal Investigator — Department of Geriatrics, Aarhus University Hospital, Denmark; Else Marie Damsgaard, MD, DMSc, Study Director — Department of Geriatrics, Aarhus University Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department of Geriatrics, Aarhus University Hospital, Aarhus
  - Rehabilitation Unit Vikaergaarden and Thorsgaarden, Aarhus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zintchouk D, Gregersen M, Lauritzen T, Damsgaard EM. Geriatrician-performed comprehensive geriatric care in older adults referred to an outpatient community rehabilitation unit: A randomized controlled trial. Eur J Intern Med. 2018 May;51:18-24. doi: 10.1016/j.ejim.2018.01.022. Epub 2018 Feb 1. PMID 29395938